CLINICAL TRIAL: NCT06014502
Title: A Phase 1a/1b, Open-label, Dose-escalation, and Dose-expansion Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Anti-tumor Activity of IMGS-001 in Patients With Relapsed or Refractory Advanced Solid Tumors
Brief Title: Study to Evaluate IMGS-001 Treatment in Patients With Relapsed or Refractory Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: ImmunoGenesis (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: IMGS-001-011
Record Dates: First submitted 2023-08-17; First posted 2023-08-28 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Solid Tumor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (6):
- Phase 1a Solid Tumors (Experimental): IMGS-001 will be administered in escalating doses, with a starting dose of 0.3 mg/kg every 2 weeks escalating up to a maximum dose of 20 mg/kg.
  Interventions: Drug: IMGS-001
- Phase 1b Ovarian Cancer (Experimental): IMGS-001 will be administered every 2 weeks at the highest of the two doses of IMGS-001 that were selected for further evaluation in Phase 1a. Based on meeting minimum prespecified efficacy criteria, additional subjects may be enrolled and randomly assigned (1:1) to receive either the higher dose (Arm A) or a lower dose (Arm B) selected from Phase 1a.
  Interventions: Drug: IMGS-001
- Phase 1b Colorectal Cancer (Microsatellite Stable; PD-L1 Positive [CPS ≥ 5 or TPS ≥ 5%]) (Experimental): IMGS-001 will be administered every 2 weeks at the highest of the two doses of IMGS-001 that were selected for further evaluation in Phase 1a. Based on meeting minimum prespecified efficacy criteria, additional subjects may be enrolled and randomly assigned (1:1) to receive either the higher dose (Arm A) or a lower dose (Arm B) selected from Phase 1a.
  Interventions: Drug: IMGS-001
- Phase 1b Non-small Cell Lung Cancer (EGFR Wild-type) (Experimental): IMGS-001 will be administered every 2 weeks at the highest of the two doses of IMGS-001 that were selected for further evaluation in Phase 1a. Based on meeting minimum prespecified efficacy criteria, additional subjects may be enrolled and randomly assigned (1:1) to receive either the higher dose (Arm A) or a lower dose (Arm B) selected from Phase 1a.
  Interventions: Drug: IMGS-001
- Phase 1b Nasopharyngeal Cancer (Experimental): IMGS-001 will be administered every 2 weeks at the highest of the two doses of IMGS-001 that were selected for further evaluation in Phase 1a. Based on meeting minimum prespecified efficacy criteria, additional subjects may be enrolled and randomly assigned (1:1) to receive either the higher dose (Arm A) or a lower dose (Arm B) selected from Phase 1a.
  Interventions: Drug: IMGS-001
- Phase 1b Head and Neck/Cervical Cancer (HPV positive) (Experimental): IMGS-001 will be administered every 2 weeks at the highest of the two doses of IMGS-001 that were selected for further evaluation in Phase 1a. Based on meeting minimum prespecified efficacy criteria, additional subjects may be enrolled and randomly assigned (1:1) to receive either the higher dose (Arm A) or a lower dose (Arm B) selected from Phase 1a.
  Interventions: Drug: IMGS-001

INTERVENTIONS:
Drug: IMGS-001 — Every 2 weeks

SUMMARY:
The purpose of this Phase 1a/1b clinical trial is to test the safety of an investigational drug called IMGS-001 and to determine how well it can work in treating patients with advanced solid tumors that have come back or are not improving after receiving other drugs that are commonly used for their cancer. Phase 1a (Part 1) will test the safety of five different doses of IMGS-001 to use in further studies. Patients with cancer that have advanced or spread to other parts of the body following treatment with other available therapies will be treated in Part 1. Phase 1b (Part 2) will test two doses of IMGS-001 identified in Part 1 to further determine the safety and potential effectiveness in select cancer types.

DETAILED DESCRIPTION:
Part 1 is a Phase 1a, first-in-human, open-label dose-escalation study to determine the safety, tolerability, and maximum tolerated dose (MTD) of IMGS-001. The safety, tolerability, PK parameters, and preliminary antitumor activity of IMGS-001 will be assessed in adult patients with advanced solid tumors refractory to appropriate standard of care (SOC) treatments.

Based on the MTD and other information (e.g., tolerability, PK, PD, target engagement), two doses of IMGS-001 will be selected for further evaluation. Additional subjects will be backfilled until at least 10 evaluable subjects have been treated with each of these doses. Approximately 25 total subjects will be enrolled in Phase 1a.

Part 2 is a Phase 1b, open-label, dose-expansion study of five prespecified tumor cohorts to assess preliminary antitumor activity of IMGS-001 in patients that are refractory or intolerant to other appropriate prior standard therapies. Initially, up to 10 subjects in each of the following cohorts will be treated:

Cohort 1: Ovarian cancer; Cohort 2: Colorectal cancer (microsatellite stable; PD-L1 positive [CPS ≥ 5 or TPS ≥ 5%]); Cohort 3: Non-small cell lung cancer (EGFR wild-type); Cohort 4: Nasopharyngeal cancer; Cohort 5: Head and neck/cervical (HPV positive).

Each cohort will be assessed to meet efficacy criteria to continue into a randomized dose-optimization. Within each cohort that meets prespecified efficacy criteria, the expanded cohorts will have randomly assigned (1:1) subjects to receive one of two doses used in the Phase 1a. Within each Arm, 20 eligible subjects will be treated with the assigned dose of IMGS-001.

ELIGIBILITY:
Inclusion Criteria:

* Part 1 Dose-escalation: Patients must have histologically confirmed locally advanced, or metastatic solid tumors who have progressed after receiving appropriate lines of standard therapy known to potentially confer clinical benefit.
* Part 2 Dose-expansion: Patients must have histologically confirmed locally advanced, or metastatic cancer in one of the following pre-specified tumor types and meet tumor-specific criteria:

  1. Ovarian: Failed or intolerant to prior lines of appropriate SOC chemotherapy and targeted therapy regimens. Must be naïve to treatment with PD-1 and PD-L1 targeting agents.
  2. Colorectal (microsatellite stable; PD-L1 positive [CPS ≥ 5 or TPS ≥ 5%]): Failed or intolerant to prior lines of appropriate SOC chemotherapy and targeted therapy regimens. Must be naïve to treatment with PD-1 and PD-L1 targeting agents.
  3. Non-small cell lung (EGFR wild-type): Failed or intolerant to prior lines of appropriate SOC chemotherapy and targeted therapy regimens. Failed, did not respond, or intolerant to prior immune checkpoint therapy (e.g., anti-PD-1).
  4. Nasopharyngeal: Failed or intolerant to prior lines of appropriate SOC chemotherapy and targeted therapy regimens. Failed, did not respond, or intolerant to prior immune checkpoint therapy (e.g., anti-PD-L1).
  5. Head and neck/cervical (HPV positive): Failed or intolerant to prior lines of appropriate SOC chemotherapy and targeted therapy regimens. Failed, did not respond, or intolerant to prior immune checkpoint therapy (e.g., anti-PD-L1).
* Prostate cancer patients enrolled in Part 1 dose escalation must continue ongoing androgen deprivation therapy with a gonadotropin-releasing hormone (GnRH) analog or have undergone a bilateral orchiectomy (surgical or medical castration) and must have a serum testosterone ≤1.73 nmol/L (50 ng/dL) at screening.
* Patients eligible to enroll in cohorts with prior immune checkpoint therapy must meet the following criteria:

  1. Received at least 2 doses of an approved or investigational anti PD-1 or anti-PD-L1 inhibitor.
  2. Last dose of therapy must have been ≥ 28 days prior to Cycle 1 Day 1.
  3. Eligible patients include those patients treated with anti PD-1/anti PD-L1 drugs who have progressed following response to prior therapy, and those that have failed to demonstrate any response to prior therapy.
* Colorectal patients participating in Part 2 (Phase 1b) must have confirmed PD-L1 positive expression (CPS ≥ 5 or TPS ≥ 5%) using local laboratory results based on prior results obtained within 6 months of baseline, expression testing done on archived tissue within 6 calendar months of baseline, or fresh biopsy.
* Male or female ≥ 18 years of age.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-1.
* Life expectancy > 3 months.
* At least one measurable lesion as defined by RECIST 1.1.

  a. A lesion that was previously irradiated may be considered a target lesion only if it is measurable per RECIST 1.1, has documented progression, and is clearly defined.
* Patients must have a non-target lesion that can be biopsied. If a patient only has one target lesion (and no non-target lesions) the target lesion used for biopsy must be ≥ 2 cm in longest diameter. Eligible subjects for biopsy must be clinically appropriate, including specimens attainable and on appropriate subjects without presenting high risk of major complications. Subjects who are unable to undergo a biopsy at screening must submit archival tumor tissue retrieved within the last 6 months.
* Patients must have adequate bone marrow and organ function as defined by:

  1. Absolute neutrophil count (ANC) ≥ 1.5×10^9/L.
  2. Platelet count of ≥ 100.0×10^9/L.
  3. Hemoglobin of ≥ 9.0 g/dL.
  4. Creatinine clearance ≥ 30 mL/min.
  5. Liver function test: AST (SGOT) and ALT (SGPT) ≤ 2.5 times the institutional ULN.
  6. Total bilirubin: ≤ 1.5 x ULN.

Exclusion Criteria:

* Receipt of any investigational or conventional anti-cancer drug/therapy within 21 days of Cycle 1 Day 1.
* Current or prior use of immunosuppressive medication within 14 days of Cycle 1 Day 1. Inhaled and intranasal corticosteroids are allowed.
* Current or prior use of interleukin-2, interferon, or other immunotherapy medication within 28 days of Cycle 1 Day 1.
* Live vaccine within 28 days prior to Cycle 1 Day 1.
* Any toxicity from prior standard therapy that has not resolved to ≤ Grade 1 or baseline per National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 5.0 at the time of consent. Alopecia is an exception. Any patients with irreversible Grade 1 or Grade 2 toxicities that are considered stable may be enrolled after discussion with the Medical Monitor.
* Prior anti-PD-1 or anti-PD-L1-related Grade 3 or Grade 4 toxicity resulting in treatment discontinuation of the drug.
* Secondary malignancy other than the target malignancy to be investigated in this trial within the last 2 years.
* History of myocardial infarction, ischemic heart disease, symptomatic congestive heart failure (New York Heart Association (NYHA) Class III IV), or significant cardiac arrhythmias within 3 months of study enrollment.
* Arterial or venous thrombotic or embolic events such as cerebrovascular accident (including transient ischemic attacks) or pulmonary embolism within 3 months of study enrollment.
* History of acute diverticulitis, intra-abdominal abscess, gastrointestinal (GI) obstruction, abdominal carcinomatosis, bowel perforation, or other known risk factors for bowel perforation.
* Active, uncontrolled, or prior documented autoimmune disorders including but not limited to inflammatory bowel disease (including Crohn's disease and ulcerative colitis), rheumatoid arthritis, systemic sclerosis (scleroderma), Systemic Lupus Erythematosus, or autoimmune vasculitis (e.g., Wegener's Granulomatosis). Alopecia, vitiligo, celiac disease controlled by diet, and chronic skin conditions not requiring systemic therapy/immunosuppressive treatment is permitted.
* Uncontrolled intercurrent illness, including active infection requiring systemic therapy, uncontrolled hypertension (> 150/90mm Hg despite optimal medical management), uncontrolled asthma, psychiatric illness/social situations, substance abuse, or other underlying medical conditions that would limit compliance with study requirements, obscure the interpretation of AEs, substantially increase the risk of developing AEs, or make the administration of study treatment hazardous.
* Active human immunodeficiency virus (HIV) infection (Exception: patients with well-controlled HIV [e.g., CD4 ≥ 350 cells/uL and undetectable viral load] who have been on an effective [drug, dosage, and schedule associated with reduction and control of the viral load] antiretroviral therapy [ART] for ≥ 4 weeks are eligible). Patients with a history of acquired immunodeficiency syndrome (AIDS)-defining opportunistic infections in the last 12 months are not eligible.
* Active or chronic hepatitis B virus (HBV) or hepatitis C virus (HCV) infection. Patients with a history of HCV infection must have completed curative antiviral treatment and must have a viral load below the limit of quantification. A patient who is HCV antibody (Ab) positive but HCV RNA negative due to prior treatment or natural resolution is eligible.
* History of solid organ transplantation.
* Newly diagnosed, uncontrolled, and/or untreated cancer-related central nervous system disease. Patients with treated brain metastases that are radiographically or clinically stable for at least 28 days after therapy and have no evidence of cavitation or hemorrhage in the brain lesion(s) are eligible if they are asymptomatic and do not require corticosteroids (the patient must have discontinued steroids at least 14 days prior to Cycle 1 Day 1).
* Major surgery, open biopsy, or significant traumatic injury within 28 days of Cycle 1 Day 1, or still recovering from prior surgery. Port placement and other local procedures are allowed if completed at least 48 hours prior to Cycle 1 Day 1.
* Abnormal pulmonary function within the previous 6 months prior to Cycle 1 Day 1, including history of or active pneumonitis, interstitial lung disease requiring the use of steroids, idiopathic pulmonary fibrosis, recurrent pleural effusion (including malignant origin), severe dyspnea at rest or requiring supplementary oxygen therapy.
* Patients who have experienced any infusion related reaction Grade 3 or higher from prior therapy per NCI CTCAE version 5.0

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Estimated)
Dates: Start 2023-09-07 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Phase 1a- Safety and tolerability of IMGS-001 by dose-limiting toxicities and adverse events | 21 days
  Frequency and severity of dose limiting toxicities and adverse events
Phase 1b- Recommended Phase 2 dose (RP2D) of IMGS-001 for specified tumor-specific cohorts as a pharmacologically optimal dose (POD) | 12 months
  RP2D will be defined by pooling all available PK, PD, target engagement, efficacy, safety, and tolerability data from Part 1 and Part 2

SECONDARY OUTCOMES:
Phase 1a- Maximum tolerable dose (MTD) of IMGS-001 | 12 months
Pharmacokinetics (PK) of IMGS-001 by terminal half life (t1/2) | 12 months
Pharmacokinetics of IMGS-001 by Area Under the Curve (AUC) | 12 months
Pharmacokinetics of IMGS-001 by Maximum Observed Concentration (Cmax) | 12 months
Pharmacokinetics of IMGS-001 by Minimum Observed Concentration (Cmin) | 12 months
Potential immunogenicity of IMGS-001 by measurement of positive anti-drug antibody (ADA) levels | 12 months
Efficacy of IMGS-001 by Objective Response Rate (ORR) via RECIST 1.1 and iRECIST | 12 months
Efficacy of IMGS-001 by Progression Free Survival (PFS) | 12 months
Efficacy of IMGS-001 by Duration of Response (DOR) | 12 months
Efficacy of IMGS-001 by Clinical Benefit Rate (CBR) | 12 months
Phase 1b- Safety and tolerability of IMGS-001 by frequency and severity of Adverse Events | 12 months

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Banner MD Anderson Cancer Center, Gilbert, Arizona
  - Sarcoma Oncology Center, Santa Monica, California
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - MD Anderson Cancer Center, Houston, Texas
  - NEXT Dallas, Irving, Texas

IPD SHARING:
Plan to Share IPD: No